CLINICAL TRIAL: NCT07079826
Title: Sparrow Link Device for Opioid Withdrawal Management at UPMC Presbyterian With the Substance Treatment and Recovery Service (STARS; Formerly Addiction Medicine Consult Service)
Brief Title: Sparrow Link Neuromodulation Device for Opioid Withdrawal Management in Hospitalized Adults With Opioid Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Payel Roy (Other)
Collaborators: UPMC Ladies Hospital Aid Society (Unknown)
Responsible Party: Sponsor-Investigator, Payel Roy, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY24050080
Record Dates: First submitted 2025-06-20; First posted 2025-07-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Opioid Withdrawal; Opioid Use Disorder (OUD)
Keywords: transcutaneous auricular neurostimulation; Sparrow Link; tAN; vagus nerve stimulation; trigeminal nerve stimulation; neuromodulation; Clinical Opiate Withdrawal Scale; opioid craving; inpatient addiction care; withdrawal management; Addiction Medicine; anxiety; depression
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tAN + Standard Care (Active Comparator): Active tAN stimulation in addition to standard of care for opioid withdrawal management
  Interventions: Device: Sparrow Link (Active tAN)
- Sham tAN + Standard Care (Sham Comparator): Sham tAN stimulation in addition to standard of care for opioid withdrawal management
  Interventions: Device: Sparrow Link (Sham tAN)

INTERVENTIONS:
Device: Sparrow Link (Active tAN) — Participants will receive the Sparrow Link device with active transcutaneous auricular neurostimulation (tAN) in addition to standard hospital-based opioid withdrawal management. Standard care may include pharmacologic treatments such as methadone, buprenorphine, full agonist opioids (e.g., oxycodone), and non-opioid medications, as clinically indicated.
  Arms: Active tAN + Standard Care
Device: Sparrow Link (Sham tAN) — Participants will receive the Sparrow Link device with sham (non-active) stimulation in addition to standard hospital-based opioid withdrawal management. Standard care may include pharmacologic treatments such as methadone, buprenorphine, full agonist opioids (e.g., oxycodone), and non-opioid medications, as clinically indicated.
  Arms: Sham tAN + Standard Care

SUMMARY:
This study is evaluating the Sparrow Link, a wearable device that delivers gentle electrical signals to nerves in the outer ear (a technique known as transcutaneous auricular neurostimulation, or tAN). The goal is to assess whether the device is feasible to use, acceptable to patients, and may help reduce opioid withdrawal symptoms in hospitalized adults being treated for opioid use disorder (OUD). Participants will be randomly assigned to receive either the active device or a sham (inactive) version. Neither participants nor their clinical teams will know which version is used. All participants will continue receiving standard hospital care for opioid withdrawal. Researchers will collect information on how long participants use the device, whether they stop using it early, and changes in withdrawal severity. The study will also examine pain, craving, mood, anxiety, heart rate variability, and opioid use during hospitalization.

DETAILED DESCRIPTION:
Opioid withdrawal is a major barrier to the initiation and continuation of treatment for opioid use disorder (OUD), particularly during hospitalization. Symptoms of withdrawal may lead patients to decline initiation of treatment or leave against medical advice. Neuromodulation strategies, such as transcutaneous auricular neurostimulation (tAN), are emerging as potential adjuncts to standard pharmacologic management. tAN targets cranial nerves via stimulation of the auricular branch of the vagus nerve and other nerve branches in the external ear. The Sparrow Link is a wearable tAN device intended for short-term use in clinical environments and is being evaluated in this study for its role in reducing withdrawal symptoms and enhancing the inpatient care experience.

This is a double-blind, sham-controlled, randomized pilot trial designed to evaluate the feasibility, acceptability, and preliminary effectiveness of the Sparrow Link device in hospitalized adults with OUD undergoing opioid withdrawal. The study is being conducted at UPMC Presbyterian and Montefiore hospitals with clinical oversight by the STARS (Substance Treatment and Recovery Service) addiction medicine consult team.

Eligible participants will be randomized 1:1 to receive either active or sham tAN stimulation. All participants will receive standard hospital-based opioid withdrawal management, including pharmacologic treatment as clinically indicated (e.g., methadone, buprenorphine, or full opioid agonists). The device is applied and monitored by trained research staff during daytime hours.

The study includes both implementation and effectiveness endpoints. Primary implementation outcomes include device usage consistency and early device discontinuation. The primary effectiveness outcome is change in opioid withdrawal severity, as measured by the Clinical Opiate Withdrawal Scale (COWS). The study also includes secondary measures of pain, anxiety, depressive symptoms, craving, heart rate variability, and opioid use during hospitalization. Exploratory outcomes include referral to follow-up care, intent to continue device use, and qualitative feedback from providers regarding device feasibility and integration into clinical workflow.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must meet at least ONE of the following criteria:

1. Are continuing to experience opioid withdrawal symptoms:

   1. Despite Maximal medical therapy with methadone, buprenorphine, full agonist opioids, or non-opioid medications,

      or
   2. During tapering or detox from full agonist opioids.

   OR
2. Have chosen to decline methadone or buprenorphine but still require support for withdrawal symptoms and/or pain management.

Additionally, participants must:

* Be 18 years old or older.
* Have active history of opioid use disorder.
* Have a COWS score between 5-24 (Mild-moderate opioid withdrawal), indicating residual withdrawal symptoms.
* Be able to provide informed consent.

Exclusion Criteria:

* History of or active seizure disorder.
* Presence of a cardiac device (e.g., pacemaker, defibrillator).
* Presence of a neurostimulator (e.g., deep brain stimulator, spinal cord stimulator).
* Pregnant or lactating individuals.
* COWS score ≥ 25 (Severe Withdrawal), requiring medical stabilization.
* Abnormal ear Anatomy, ear Infections, or skin Conditions at Electrode Sites, including congenital malformations, post-surgical changes, significant scarring, open wounds, or hypersensitivity.
* Active neurological disorders, such as traumatic brain injury, stroke, multiple sclerosis, or other conditions that may interfere with neurostimulation effects or autonomic regulation as assessed at the investigator's discretion.
* Severe alcohol or benzodiazepine withdrawal that is not adequately controlled with medication, per investigator discretion.
* Known or documented allergy to hydrocolloid adhesives, as evidenced in the medical record.
* Evidence of active psychosis, as documented in the medical record or reported by clinical staff.
* Non-English speakers, whose limited English proficiency precludes informed consent or meaningful participation in study assessments validated only in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-21 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Device Usage Consistency (Percentage of Expected Wear Time Achieved) | From Day 1 through the final day of device wear or early device discontinuation (up to 5 days).
  Device usage consistency is defined as the total number of hours the device was actively worn divided by the total number of hours the device was expected to be worn, multiplied by 100. Calculated using stimulation logs and staff-logged application/removal times.
Early Device Discontinuation (Percentage of Participants) | From Day 1 through the final day of device wear or early device discontinuation (up to 5 days).
  Proportion of participants who permanently discontinue device use prior to reaching protocol-defined endpoints: (1) meeting 3 of 4 clinical criteria, (2) completion of 5 study days, or (3) hospital discharge. Calculated as number discontinued divided by number who initiated use times 100.
Clinical Opiate Withdrawal Scale (COWS) | Pre-device baseline, 1-hour post-initiation, 2-hour post-initiation, and end-of-day on Day 1; then on each subsequent device wear day (Days 2-5 or until study exit), at three timepoints: pre-device, 1-hour post-device, and end-of-day (up to 5 days total)
  Opioid withdrawal severity using the Clinical Opiate Withdrawal Scale (COWS), an 11-item clinician-rated tool with scores ranging from 0-48. The primary outcome is change from pre-device baseline to 1-hour post-device placement. Higher COWS scores indicate greater opioid withdrawal severity.

SECONDARY OUTCOMES:
Early Device Refusal Rate (Percentage) | Day 1
  Proportion of randomized participants who decline to initiate device use after allocation.
Device Discomfort Reported (Percentage) | From Day 1 through the final day of device wear or early device discontinuation (up to 5 days).
  Proportion of participants reporting discomfort or physical side effects while wearing the device, regardless of discontinuation.
Technical Issue Rate (Percentage) | From Day 1 through the final day of device wear or early device discontinuation (up to 5 days).
  Proportion of participants in the active arm who experience one or more technical issues (e.g., stimulation interruption, electrode detachment, app malfunction).
Referral to Follow-Up Care Rate (Percentage) | Through study completion, an average of 5 days
  Proportion of participants discharged (planned or unplanned) with a documented referral to outpatient treatment (Medications for Opioid Use Disorder, Medication-Assisted Treatment, or other follow-up addiction treatment.)
Intent to Engage in Care Rate (Percentage) | Assessed once at the final study exit interview (interview may occur for up to 5 days post-discharge).
  Proportion of participants who express intent to attend follow-up treatment post-discharge.
Post-Discharge Engagement Composite (Percentage) | Assessed once at the final study exit interview (interview may occur for up to 5 days post-discharge).
  Composite outcome defined as presence of either: (a) documented referral or (b) participant-reported intent to engage in care.
Desire to Continue Device Use (Percentage) - Active Arm Only | Assessed once at the final study exit interview (interview may occur for up to 5 days post-discharge).
  Proportion of active-arm participants expressing desire to use the device again in the future for opioid withdrawal management.

OTHER OUTCOMES:
Subjective Opioid Withdrawal Scale (SOWS) | Pre-device baseline, 1-hour post-device, 2- hour post device, and end-of-day on Day 1; then pre-device, 1- hour post-device, end-of-day on Days 2-5 or until study exit (up to 5 days).
  16-item participant-reported scale (0-64) assessing withdrawal severity.
Numeric Pain Rating Scale (NPRS) | Pre-device baseline, 1-hour post-device, 2- hour post device, and end-of-day on Day 1; then pre-device, 1- hour post-device, end-of-day on Days 2-5 or until study exit (up to 5 days).
  Participant-reported pain severity (0-10).
Opioid Craving Scale (OCS-3) | Pre-device baseline, 1-hour post-device, 2- hour post device, and end-of-day on Day 1; then pre-device, 1- hour post-device, end-of-day on Days 2-5 or until study exit (up to 5 days).
  3-item scale measuring craving frequency, intensity, and situational response (0-30 total).
STAI-S (State-Trait Anxiety Inventory - State) | Pre-device baseline, 1-hour post-device, 2- hour post device, and end-of-day on Day 1; then pre-device, 1- hour post-device, end-of-day on Days 2-5 or until study exit (up to 5 days).
  20-item scale measuring state anxiety (range 20-80).
MADRS (Montgomery-Åsberg Depression Rating Scale) | Assessed at baseline and final study assessment (Day 5 or early discontinuation).
  Clinician-rated 10-item depression severity scale (0-60 total).
Heart Rate Variability (HRV) | Pre-device baseline, 1-hour post-device, 2- hour post device, and end-of-day on Day 1; then pre-device, 1- hour post-device, end-of-day on Days 2-5 or until study exit (up to 5 days).
  RMSSD from 5-min resting ECG using wrist wearable; reflects autonomic tone.
Mean MME per 24-Hour Period Anchored to Device Wear (Normalized) | Day 0 through up to Day 5
  Mean morphine milligram equivalents (MME) administered per 24-hour window anchored to device placement time. Normalized using: (Total MME divided by hours covered) times 24.

CONTACTS AND LOCATIONS:
Overall Officials: Payel J Roy, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) from this early-phase feasibility study will not be shared due to participant confidentiality concerns, consent limitations, and the exploratory nature of the trial. Given the small sample size and potential re-identifiability of participants, especially within a high-risk inpatient population, sharing IPD could pose privacy risks. Additionally, the consent form does not explicitly authorize future data sharing, and the study's non-powered design limits generalizability of individual-level findings.

REFERENCES:
- See also: Study device link — https://www.sparkbiomedical.com/research/sparrow-link